CLINICAL TRIAL: NCT03486873
Title: A Multicenter, Open-label, Phase 3 Study to Evaluate the Long-term Safety and Efficacy in Participants Who Are Currently on Treatment or in Follow-up in Studies That Include Pembrolizumab
Brief Title: Long-term Safety and Efficacy Extension Study for Participants With Advanced Tumors Who Are Currently on Treatment or in Follow-up in a Pembrolizumab (MK-3475) Study (MK-3475-587/KEYNOTE-587)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-587; MK-3475-587 (Other: MSD); KEYNOTE-587 (Other: MSD); 195006 (Registry Identifier: JAPIC-CTI); PHRR210209-002881 (Registry Identifier: PHRR); 2022-501254-10-00 (Registry Identifier: EU CT); jRCT2080224921 (Other: jRCT); U1111-1274-2274 (Registry Identifier: UTN); 2017-004417-42 (EudraCT Number)
Record Dates: First submitted 2018-03-29; First posted 2018-04-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumors; Hematologic Malignancies
Keywords: PD1; PD-1; PDL1; PD-L1
MeSH Terms: conditions — Hematologic Neoplasms | interventions — pembrolizumab; Standard of Care; lenvatinib; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Pembrolizumab 200 mg (Experimental): Participants receive pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 administrations or more for First Course participants and up to 17 administrations for Second Course participants.
  Interventions: Drug: Pembrolizumab
- Pembrolizumab 400 mg (Experimental): Participants receive pembrolizumab 400 mg via intravenous (IV) infusion on Day 1 of each 6-week cycle for up to 17 administrations or more for First Course participants and up to 8 administrations for Second Course participants.
  Interventions: Drug: Pembrolizumab
- Pembrolizumab 200 mg + SOC: Per Parent Study) (Experimental): Participants receive pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle PLUS standard of care (SOC) treatment (or per parent study if there is no SOC) for up to 35 administrations or more for First Course participants and up to 17 administrations for Second Course participants. Participants receiving a pembrolizumab-based combination treatment will receive the dose regimen of the combination drug(s) which is recommended per SOC or was used in the parent study protocol if there is no SOC recommendation.
  Interventions: Drug: Pembrolizumab; Drug: Standard of Care (SOC)
- Pembrolizumab 400 mg + SOC (Per Parent Study) (Experimental): Participants receive pembrolizumab 400 mg via IV infusion on Day 1 of each 6-week cycle PLUS SOC treatment (or per parent study if there is no SOC) for up to 17 administrations or more for First Course participants and up to 8 administrations for Second Course participants. Participants receiving a pembrolizumab-based combination treatment will receive the dose regimen of the combination drug(s) which is recommended per SOC or was used in the parent study protocol if there is no SOC recommendation.
  Interventions: Drug: Pembrolizumab; Drug: Standard of Care (SOC)
- SOC (Per Parent Study) (Active Comparator): Participants receive the dose matched non-pembrolizumab SOC treatment (e.g. chemotherapy) they were receiving as per parent study protocol.
  Interventions: Drug: Standard of Care (SOC)
- Lenvatinib 20 mg (Experimental): Participants with body weight (BW)>60kg receive Lenvatinib 20mg orally once daily on a 21 or 42 day cycle. It is taken 0-4 hours after completion of pembrolizumabd administration in the clinic on cycle 1 day 1(C1D1), C2D1, C3D1, etc. Taken at home on all other days.
  Interventions: Drug: Lenvatinib
- Lenvatinib 24 mg (Experimental): Participants with body weight (BW)>60 kg receive Lenvatinib 24 mg orally once daily on a 21 or 42 day cycle. It is taken 0-4 hours after completion of pembrolizumabd administration in the clinic on cycle 1 day 1(C1D1), C2D1, C3D1, etc. Taken at home on all other days.
  Interventions: Drug: Lenvatinib
- Lenvatinib 12 mg (Experimental): Participants with body weight (BW)>60 kg receive Lenvatinib 12 mg orally once daily on a 21 or 42 day cycle. It is taken 0-4 hours after completion of pembrolizumabd administration in the clinic on cycle 1 day 1(C1D1), C2D1, C3D1, etc. Taken at home on all other days.
  Interventions: Drug: Lenvatinib
- Lenvatinib 8 mg (Experimental): Participants with body weight (BW)<60 kg receive Lenvatinib 8 mg orally once daily on a 21 or 42 day cycle. It is taken 0-4 hours after completion of pembrolizumabd administration in the clinic on cycle 1 day 1(C1D1), C2D1, C3D1, etc. Taken at home on all other days.
  Interventions: Drug: Lenvatinib
- Lenvatinib 2mg (Experimental): Participants with body weight (BW)<60 kg receive Lenvatinib 2 mg orally once daily on a 21 or 42 day cycle. It is taken 0-4 hours after completion of pembrolizumab administration in the clinic on cycle 1 day 1(C1D1), C2D1, C3D1, etc. Taken at home on all other days.
  Interventions: Drug: Lenvatinib
- Olaparib 300mg (Experimental): Participants receive Olaparib 300 mg orally twice daily (BID) until disease progression or toxicity prohibits its administration.
  Interventions: Drug: Olaparib
- Olaparib 250mg (Experimental): Participants receive Olaparib 250 mg orally twice daily (BID) until disease progression or toxicity prohibits its administration.
  Interventions: Drug: Olaparib
- Olaparib 100mg (Experimental): Participants receive Olaparib 100 mg orally twice daily (BID) until disease progression or toxicity prohibits its administration.
  Interventions: Drug: Olaparib
- MK-4280 800mg (Experimental): Participants receive MK-4280 800mg as IV infusion every 3 weeks (Q3W) and may continue study therapy until study treatment completion or may transition to pembrolizumab to complete their treatment.
  Interventions: Drug: MK-4280
- MK-4280A (Experimental): Participants receive MK-4280A (800mg favezelimab + 200mg pembrolizumab) as IV infusion every 3 weeks (Q3W) and may continue study therapy until study treatment completion or may transition to pembrolizumab to complete their treatment.
  Interventions: Biological: MK-4280A

INTERVENTIONS:
Drug: Pembrolizumab — 200 or 400 mg IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab 200 mg; Pembrolizumab 200 mg + SOC: Per Parent Study); Pembrolizumab 400 mg; Pembrolizumab 400 mg + SOC (Per Parent Study)
Drug: Standard of Care (SOC) — IV infusion or oral tablets
  Arms: Pembrolizumab 200 mg + SOC: Per Parent Study); Pembrolizumab 400 mg + SOC (Per Parent Study); SOC (Per Parent Study)
Drug: Lenvatinib — Oral capsules
  Arms: Lenvatinib 12 mg; Lenvatinib 20 mg; Lenvatinib 24 mg; Lenvatinib 2mg; Lenvatinib 8 mg
Drug: Olaparib — 300mg or 250mg or 100mg oral tablers
  Other Names: Lynparza
  Arms: Olaparib 100mg; Olaparib 250mg; Olaparib 300mg
Drug: MK-4280 — IV Infusion
  Other Names: Favezelimab
  Arms: MK-4280 800mg
Biological: MK-4280A — 800mg favezelimab + 200mg pembrolizumab IV Infusion
  Arms: MK-4280A

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of pembrolizumab (MK-3475) in participants from previous Merck pembrolizumab-based parent studies who transition into this extension study.

This study will consist of three phases: 1) First Course Phase, 2) Survival Follow-up Phase or 3) Second Course Phase. Each participant will transition to this extension study in one of the following three phases, depending on the study phase they were in at the completion of the parent study. Participants who were in the First Course Phase of study treatment with pembrolizumab or lenvatinib in their parent study will enter the First Course Phase of this study and complete up to 35 doses or more every 3 weeks (Q3W) or 17 doses or more every 6 weeks (Q6W) of study treatment with pembrolizumab or a pembrolizumab-based combination or lenvatinib according to arm assignment. Participants who were in the Follow-up Phase in the parent study (post-treatment or Survival Follow-up Phase) will enter the Survival Follow-up Phase of this study. Participants who were in the Second Course Phase in their parent study will enter Second Course Phase of this study and complete up to 17 doses Q3W or 8 doses Q6W of study treatment with pembrolizumab or a pembrolizumab-based combination according to arm assignment.

Any participant originating from a parent trial where crossover to pembrolizumab was permitted upon disease progression may be eligible for 35 doses as Q3W or 17 doses Q6W of pembrolizumab (approximately 2 years), if they progress while on the control arm and pembrolizumab is approved for the indication in the country where the potential eligible crossover participant is being evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Treated on the parent pembrolizumab studies established by the Sponsor as MK-3475-587 ready.
* Currently receiving pembrolizumab, pembrolizumab based combinations or lenvatinib from parent studies or in a follow-up phase.

Additional eligibility criteria for participants who enter Second Course Phase once they are enrolled on MK-3475-587:

* Has not received any anticancer systemic treatment since the last dose of pembrolizumab or a pembrolizumab-based combination in First Course Phase.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Demonstrates adequate organ function.
* Have resolution of any toxic effect(s) of First Course Phase trial treatment with pembrolizumab or a pembrolizumab-based combination to Grade 1 or less (except alopecia) before trial treatment in Second Course Phase is started. If participant received major surgery or radiation therapy of >30 Gray (Gy), they must have recovered from the toxicity and/or complications of the intervention.
* A female participant is eligible to enroll if she is not pregnant, not breastfeeding, and ≥1 of the following conditions applies: A woman of childbearing potential (WOCBP) who agrees to use contraception during the study treatment period and for ≥120 days (corresponding to time needed to eliminate any study combination treatment(s) plus 30 days (a menstruation cycle) for study treatments with risk of genotoxicity.

Additional eligibility criteria for participants who enter dosing with Lenvatinib:

* Adequately controlled blood pressure (BP) to <150/90 mmHg, with or without antihypertensive medications.
* For male agrees to be abstinent from penile-vaginal intercourse OR agrees to use a highly effective contraceptive method while receiving study drug and for 7 days after the last dose of lenvatinib.
* Is female and not pregnant/breastfeeding and at least one of the following applies during the study and for ≥4 days after: is not a woman of childbearing potential (WOCBP), is a WOCBP and uses highly effective contraception (low user dependency method OR a user dependent hormonal method in combination with a barrier method) or is a WOCBP who is abstinent from heterosexual intercourse.

Exclusion Criteria:

-There are no exclusion criteria to participate in MK-3475-587.

Participants are excluded from entering Second Course trial treatment once they are enrolled on MK-3475-587 if any of the following criteria applies:

* Has severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients.
* Has received a live vaccine within 30 days prior to the first dose of Second Course Phase trial treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the Cycle 1 Day 1 of Second Course Phase.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include early stage cancers (carcinoma in situ or Stage 1) treated with curative intent, melanoma (non-ulcerated, thin primary), basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer, or in situ breast cancer that has undergone potentially curative therapy.
* Has known active central nervous system metastases and/or carcinomatous meningitis.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis. Note: Participants that experienced pneumonitis during First Course that did not meet the criteria for permanent discontinuation are eligible.
* Non-small cell lung cancer (NSCLC) participants only: Has interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has a known history of or is positive for hepatitis B or hepatitis C. For parent studies where inclusion of participants with hepatitis was permitted, MK-3475-587 will follow the parent study eligibility criteria for hepatitis.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the Second Course Phase eligibility Visit through 120 days after the last dose of study treatment.
* Has severe cardiovascular disease, i.e., arrhythmias, requiring chronic treatment, congestive heart failure (New York Heart Association Class III or IV) or symptomatic ischemic heart disease.
* Has hepatic decompensation (Child-Pugh score >6 [class B and C]).
* Has uncontrolled thyroid dysfunction.
* Has uncontrolled diabetes mellitus.
* Has had an allogeneic tissue/solid organ transplant.
* Has a known history of active tuberculosis (TB; Bacillus tuberculosis).

Additional exclusion criteria for participants who enter dosing with Lenvatinib:

* Has had major surgery within 3 weeks prior to first dose of study intervention(s).
* Has preexisting ≥Grade 3 gastrointestinal or non-gastrointestinal fistula.
* Has urine protein ≥1 g/24 hours.
* Has LVEF below the institutional (or local laboratory) normal range, as determined by multigated acquisition scan (MUGA) or echocardiogram (ECHO).
* Has radiographic evidence of encasement or invasion of a major blood vessel, or of intratumoral cavitation.
* Prolongation of QT intervals corrected for heart rate using Fridericia's (cube root) correction (QTcF) interval to >480 ms.
* Has clinically significant cardiovascular disease within 12 months from first dose of study intervention, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability.
* Gastrointestinal malabsorption or any other condition that might affect the absorption of lenvatinib.
* Active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug.
* Has a history of any contraindication or has a severe hypersensitivity to any components of lenvatinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2018-08-21 (Actual); Primary Completion 2043-08-04 (Estimated); Study Completion 2043-08-04 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 10 years
  OS is defined as the time from randomization or start of study treatment for non-randomized participants (on the parent study) to death due to any cause. Participants without documented death at the time of analysis will be censored at the date of the last known to be alive.

SECONDARY OUTCOMES:
Modified Progression Free Survival (PFS) Per Evaluation Criteria Used in the Parent Trial | Up to approximately 10 years
  Modified PFS is defined as the time from randomization or start of study treatment for nonrandomized participants (on the parent study or this study) to the first documented disease progression per the evaluation criteria used in the parent study based on investigator assessment or death due to any cause, whichever occurs first. The censoring rule is modified that participants without modified PFS events at the time of the analysis will be censored at the date of last known to be alive.
Modified Event Free Survival (EFS) Per Evaluation Criteria Used in the Parent Trial | Up to approximately 10 years
  Modified EFS is defined as the time from randomization to disease progression that precludes surgery, local or distant recurrence, or death due to any cause, whichever occurs first. The censoring rule is modified that participants without documented modified EFS events at the time of the analysis will be censored at the date of last known to be alive.
Number of Participants Who Experience Serious Adverse Events (SAEs) | Up to approximately 42 months (Up to 90 days after last dose of study treatment)
  A SAE is defined as any untoward medical occurrence that, at any dose: Results in death, Is life-threatening, Requires inpatient hospitalization or prolongation of existing hospitalization, Results in persistent or significant disability/incapacity or Is a congenital anomaly/birth defect. The number of participants who experience a SAE in this study will be presented.
Number of Participants Who Experience Adverse Events of Special Interest (AEOSI) | Up to approximately 40 months (Up to 30 days after last dose of study treatment)
  AEOSI for this study include selected preferred terms from Medical Dictionary for Regulatory Activities (MedDRA) version 20.1 for the following higher-level terms: Pneumonitis, Colitis, Hepatitis, Nephritis, Adrenal Insufficiency, Hypophysitis, Hyperthyroidism, Hypothyroidism, Thyroiditis, Type 1 Diabetes Mellitus, Severe Skin Reactions Including Stevens-Johnson Syndrome (SJS) and Toxic Epidermal Necrolysis (TEN): or If grade 3 or higher, Uveitis, Pancreatitis, Myositis, Guillain-Barre Syndrome, Myocarditis, Encephalitis, Sarcoidosis, Infusion Reactions and Myasthenic Syndrome. The number of participants who experience an AEOSI in this study will be presented.
Number of Participants Who Experience Clinically Significant Adverse Events (CSAE) | Up to approximately 40 months (Up to 30 days after last dose of study treatment)
  CSAE are AEs associated with lenvatinib treatment and include selected preferred terms from the lenvatinib CSAE preferred term list document. The number of participants who experience an CSAE in this study will be presented.
Number of Participants Who Experience Events of Clinical Interest (ECI) | Up to approximately 40 months (Up to 30 days after last dose of study treatment)
  ECIs for this study include: 1) An overdose of Sponsor's product, that is not associated with clinical symptoms or abnormal laboratory results or 2) An elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) lab value that is ≥3X the upper limit of normal (ULN) and an elevated total bilirubin lab value that is ≥2X ULN and, at the same time, an alkaline phosphatase lab value that is <2X ULN, as determined by way of protocol-specified laboratory testing or unscheduled laboratory testing. The number of participants who experience an ECI in this study will be presented.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 39 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinue study treatment due to an AE will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (772):
- United States (65):
  - Arizona Cancer Center at UMC North ( Site 0018), Tucson, Arizona
  - Comprehensive Blood & Cancer Center [Bakersfield, CA] ( Site 0054), Bakersfield, California
  - California Cancer Associates for Research & Excellence ( Site 0016), Fresno, California
  - Providence Medical Foundation ( Site 0087), Fullerton, California
  - The Angeles Clinic and Research Institute ( Site 0005), Los Angeles, California
  - UCLA Hematology/Oncology - Westwood (Building 100) ( Site 0009), Los Angeles, California
  - University of California, Irvine (UCI) Health - UC Irvine Medical Center ( Site 0076), Orange, California
  - Stanford Cancer Center ( Site 0086), Palo Alto, California
  - UCSF Helen Diller Family Comprehensive Cancer Center ( Site 0004), San Francisco, California
  - Providence Saint John's Health Center ( Site 0059), Santa Monica, California
  - University of Colorado Cancer Center ( Site 0021), Aurora, Colorado
  - Yale Cancer Center ( Site 0014), New Haven, Connecticut
  - Georgetown University Medical Center ( Site 0023), Washington D.C., District of Columbia
  - Holy Cross Hospital, Michael & Dianne Bienes Comp Cancer Ctr ( Site 0022), Fort Lauderdale, Florida
  - Baptist MD Anderson Cancer Center ( Site 0083), Jacksonville, Florida
  - Mount Sinai Medical Center Comprehensive Cancer Center ( Site 0031), Miami Beach, Florida
  - Moffitt Cancer Center ( Site 0011), Tampa, Florida
  - Emory School of Medicine ( Site 0013), Atlanta, Georgia
  - Augusta University ( Site 0077), Augusta, Georgia
  - Northwest Georgia Oncology Centers PC ( Site 0061), Marietta, Georgia
  - Kaiser Permanente Moanalua Medical Center ( Site 0063), Honolulu, Hawaii
  - The University of Chicago ( Site 0020), Chicago, Illinois
  - University of Iowa Hospital and Clinics ( Site 0026), Iowa City, Iowa
  - James Graham Brown Cancer Center ( Site 0058), Louisville, Kentucky
  - Mercy Health-Paducah Cancer Center ( Site 0084), Paducah, Kentucky
  - Women's Cancer Care ( Site 0088), Covington, Louisiana
  - MedStar Franklin Square Medical Center ( Site 0046), Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins ( Site 0056), Baltimore, Maryland
  - Maryland Oncology Hematology (MOH) ( Site 8000), Columbia, Maryland
  - Massachusetts General Hospital ( Site 0041), Boston, Massachusetts
  - Dana-Farber Cancer Institute ( Site 0006), Boston, Massachusetts
  - Karmanos Cancer Institute ( Site 0047), Detroit, Michigan
  - Mayo Clinic in Rochester, Minnesota ( Site 0002), Rochester, Minnesota
  - Comprehensive Cancer Centers of Nevada ( Site 0043), Las Vegas, Nevada
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0038), Hackensack, New Jersey
  - Cancer Institute of New Jersey ( Site 0025), New Brunswick, New Jersey
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health ( Site 0032), New York, New York
  - Memorial Sloan Kettering Cancer Center ( Site 0012), New York, New York
  - White Plains Hospital-Center for Cancer Care ( Site 0069), White Plains, New York
  - WakeMed Cancer Care - Waverly Hematology & Medical Oncology ( Site 0074), Cary, North Carolina
  - University of North Carolina at Chapel Hill ( Site 0040), Chapel Hill, North Carolina
  - Levine Cancer Institute ( Site 0034), Charlotte, North Carolina
  - Duke Cancer Center ( Site 0028), Durham, North Carolina
  - Sanford Fargo Medical Center-Roger Maris Cancer Center ( Site 0065), Fargo, North Dakota
  - University Hospitals ( Site 0044), Cleveland, Ohio
  - Oklahoma Cancer Specialists and Research Institute, LLC ( Site 0082), Tulsa, Oklahoma
  - Providence Portland Medical Center ( Site 0051), Portland, Oregon
  - St. Luke's University Health Network ( Site 0017), Bethlehem, Pennsylvania
  - University of Pennsylvania ( Site 0010), Philadelphia, Pennsylvania
  - Fox Chase Cancer Center ( Site 0042), Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center ( Site 0008), Pittsburgh, Pennsylvania
  - Saint Francis Health System ( Site 0089), Greenville, South Carolina
  - Sanford Cancer Center ( Site 0066), Sioux Falls, South Dakota
  - West Cancer Center and Research Institute ( Site 0055), Germantown, Tennessee
  - Vanderbilt Health One Hundred Oaks Diagnostic ( Site 0060), Nashville, Tennessee
  - Vanderbilt Ingram Cancer Center ( Site 0015), Nashville, Tennessee
  - Texas Oncology - Central/South Texas ( Site 8001), Austin, Texas
  - Texas Oncology-Baylor Sammons Cancer Center ( Site 0062), Dallas, Texas
  - University of Texas MD Anderson Cancer Center ( Site 0007), Houston, Texas
  - South Texas Accelerated Research Therapeutics, LLC (START) ( Site 0001), San Antonio, Texas
  - University of Virginia Health System ( Site 0035), Charlottesville, Virginia
  - Bon Secours St. Francis Medical Center-Oncology Research ( Site 0075), Midlothian, Virginia
  - VCU Health Adult Outpatient Pavillion ( Site 0080), Richmond, Virginia
  - Blue Ridge Cancer Care ( Site 0067), Roanoke, Virginia
  - Fred Hutchinson Cancer Center ( Site 0024), Seattle, Washington
- Argentina (21):
  - Centro de Oncología e Investigación de Buenos Aires ( Site 1357), Berazategui, Buenos Aires
  - Centro de Educación Médica e Investigaciones clínicas "Dr. Norberto Quirno" (CEMIC) ( Site 1368), Buenos Aires., Buenos Aires
  - Fundacion Favaloro ( Site 1367), CABA, Buenos Aires
  - Derma Internacional SA ( Site 1372), CABA, Buenos Aires
  - Instituto Alexander Fleming ( Site 1364), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - IDIM - Instituto de Investigaciones Metabólicas ( Site 1362), Ciudad de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 1363), Mar del Plata, Buenos Aires
  - Instituto Médico Río Cuarto ( Site 1375), Río Cuarto, Córdoba Province
  - Clinica Viedma ( Site 1353), Viedma, Río Negro Province
  - Fundacion Estudios Clinicos ( Site 1369), Rosario, Santa Fe Province
  - Sanatorio Parque ( Site 1355), Rosario, Santa Fe Province
  - Instituto de Oncologia de Rosario ( Site 1350), Rosario, Santa Fe Province
  - Hospital Provincial del Centenario ( Site 1359), Rosario, Santa Fe Province
  - Hospital Aleman-Oncology ( Site 1351), Buenos Aires
  - Clínica Universitaria Reina Fabiola ( Site 1376), Córdoba
  - Centro Medico Privado CEMAIC ( Site 1371), Córdoba
  - Hospital Privado Universitario de Córdoba ( Site 1354), Córdoba
  - Fundación CORI para la Investigación y Prevención del Cáncer ( Site 1358), La Rioja
  - Instituto San Marcos ( Site 1366), San Juan
  - Centro Medico San Roque-Oncology ( Site 1352), San Miguel de Tucumán
  - Centro Oncologico Norte. ( Site 1370), Santiago del Estero
- Australia (30):
  - Chris OBrien Lifehouse ( Site 3003), Camperdown, New South Wales
  - Royal Prince Alfred Hospital-A.W. Morrow Gastroenterology and Liver Centre ( Site 3016), Camperdown, New South Wales
  - Liverpool Hospital-Medical Oncology ( Site 3021), Liverpool, New South Wales
  - Macquarie University ( Site 3010), Macquarie University, New South Wales
  - Mater Hospital Sydney ( Site 3007), North Sydney, New South Wales
  - Orange Hospital-Clinical Trials Unit ( Site 3027), Orange, New South Wales
  - Port Macquarie - Mid North Coast Cancer Institute-Medical Oncology ( Site 3020), Port Macquarie, New South Wales
  - Royal North Shore Hospital-Medical Oncology Clinical Trials ( Site 3025), St Leonards, New South Wales
  - Calvary Mater Newcastle ( Site 3005), Waratah, New South Wales
  - Westmead Hospital ( Site 3000), Westmead, New South Wales
  - Melanoma Institute Australia ( Site 3001), Wollstonecraft, New South Wales
  - Mater Misericordiae Limited-Medical Oncology ( Site 3019), Brisbane, Queensland
  - Gallipoli Medical Research Ltd ( Site 3011), Brisbane, Queensland
  - Royal Brisbane and Women's Hospital ( Site 3009), Herston, Queensland
  - Gold Coast University Hospital ( Site 3028), Southport, Queensland
  - Tasman Oncology Research Pty Ltd ( Site 3012), Southport, Queensland
  - Sunshine Coast University Private Hospital-Coastal Cancer Care ( Site 3032), Sunshine Coast, Queensland
  - The Townsville Hospital ( Site 3017), Townsville, Queensland
  - Princess Alexandra Hospital ( Site 3002), Woolloongabba, Queensland
  - Royal Adelaide Hospital ( Site 3014), Adelaide, South Australia
  - The Queen Elizabeth Hospital ( Site 3026), Woodville, South Australia
  - Monash Health ( Site 3015), Clayton, Victoria
  - Austin Health-Austin Hospital ( Site 3004), Heidelberg, Victoria
  - Peter MacCallum Cancer Centre-Parkville Cancer Clinical Trials Unit (PCCTU) ( Site 3008), Melbourne, Victoria
  - St Vincent's Hospital-Oncology Clinical Trials ( Site 3018), Melbourne, Victoria
  - Western Health-Sunshine & Footscray Hospitals ( Site 3023), St Albans, Victoria
  - Ballarat Oncology & Haematology Services ( Site 3022), Wendouree, Victoria
  - Fiona Stanley Hospital ( Site 3029), Murdock, Western Australia
  - Sir Charles Gairdner Hospital ( Site 3006), Nedlands, Western Australia
  - St John of God Subiaco Hospital ( Site 3013), Subiaco, Western Australia
- Austria (7):
  - Medical University of Graz ( Site 2952), Graz, Styria
  - Medizinische Universitaet Innsbruck ( Site 2951), Innsbruck, Tyrol
  - Ordensklinikum Linz GmbH Elisabethinen-Department of Pneumology ( Site 2957), Linz, Upper Austria
  - Kepler Universitätsklinikum ( Site 2955), Linz, Upper Austria
  - Uniklinikum Salzburg ( Site 2956), Salzburg
  - Medizinische Universität Wien ( Site 2953), Vienna
  - Klinik Floridsdorf-Abteilung für Innere Medizin und Pneumologie ( Site 2954), Vienna
- Belgium (10):
  - AZ Sint-Maarten ( Site 2904), Mechelen, Antwerpen
  - Institut Jules Bordet ( Site 2903), Anderlecht, Bruxelles-Capitale, Region de
  - Cliniques Universitaires de Bruxelles - CUB - Hopital Erasme ( Site 2905), Brussels, Bruxelles-Capitale, Region de
  - UZ Brussel ( Site 2900), Brussels, Bruxelles-Capitale, Region de
  - Cliniques universitaires Saint-Luc-Medical Oncology ( Site 2911), Brussels, Bruxelles-Capitale, Region de
  - AZ Maria Middelares ( Site 2908), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 2901), Leuven, Vlaams-Brabant
  - UZ Leuven - Campus Gasthuisberg ( Site 2906), Leuven, Vlaams-Brabant
  - UZ Leuven Gasthuisberg, Gynaecologie-Verloskunde ( Site 2907), Leuven, Vlaams-Brabant
  - Université Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant-Godinne - Site Godi ( Site 2909), Namur
- Brazil (28):
  - Hospital São Carlos-Oncocentro Ce ( Site 1029), Fortaleza, Ceará
  - CRIO - CENTRO REGIONAL INTEGRADO DE ONCOLOGIA-Pesquisa Clínica ( Site 1024), Fortaleza, Ceará
  - Centro de Pesquisa Clínica do Instituto do Câncer do Ceará ( Site 1016), Fortaleza, Ceará
  - Hospital Erasto Gaertner ( Site 1036), Curitiba, Paraná
  - Hospital Tacchini ( Site 1040), Bento Gonçalves, Rio Grande do Sul
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia ( Site 1008), Ijuí, Rio Grande do Sul
  - Hospital de Clínicas de Passo Fundo ( Site 1025), Passo Fundo, Rio Grande do Sul
  - Lacks - Oncologia E Hematologia ( Site 1026), Pelotas, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre ( Site 1000), Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS-Centro de Pesquisa em Oncologia ( Site 1006), Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceição ( Site 1011), Porto Alegre, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre ( Site 1035), Porto Alegree, Rio Grande do Sul
  - Clinica Viver ( Site 1021), Santa Maria, Rio Grande do Sul
  - Instituto de Oncologia Saint Gallen ( Site 1039), Ssanta Cruz Do Sul, Rio Grande do Sul
  - CEPEN - Centro de Pesquisa e Ensino em Oncologia de Santa Catarina ( Site 1034), Florianópolis, Santa Catarina
  - CEPON ( Site 1012), Florianópolis, Santa Catarina
  - Centro de Novos Tratamentos Itajai - Clinica de Neoplasias Litoral ( Site 1041), Itajaí, Santa Catarina
  - Fundação Pio XII - Hospital de Câncer de Barretos ( Site 1010), Barretos, São Paulo
  - Hospital Amaral Carvalho ( Site 1023), Jaú, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto-Centro Integrado de Pesquisa ( Site 1003), São José do Rio Preto, São Paulo
  - Clínica de Pesquisa e Centro de Estudos em Ginecologia Oncológica e Mamária LTDA ( Site 1017), São Paulo, São Paulo
  - Instituto Nacional de Câncer José Alencar Gomes da Silva - INCA ( Site 1020), Rio de Janeiro
  - Instituto de de Educação, pesquisa e Gestão em Saúde ( Site 1014), Rio de Janeiro
  - Instituto do Cancer do Estado de Sao Paulo - ICESP ( Site 1001), São Paulo
  - BP - A Beneficencia Portuguesa de São Paulo-Medical Oncology ( Site 1030), São Paulo
  - Hospital Paulistano ( Site 1033), São Paulo
  - A. C. Camargo Cancer Center ( Site 1002), São Paulo
  - Núcleo de Pesquisa Clínica da Rede São Camilo ( Site 1018), São Paulo
- Canada (19):
  - Arthur J.E. Child Comprehensive Cancer Centre ( Site 2815), Calgary, Alberta
  - Cross Cancer Institute ( Site 2804), Edmonton, Alberta
  - CancerCare Manitoba ( Site 2814), Winnipeg, Manitoba
  - Hamilton Health Sciences-Juravinski Cancer Centre ( Site 2801), Hamilton, Ontario
  - Kingston Health Sciences Centre-Kingston General Hospital Site ( Site 2808), Kingston, Ontario
  - London Health Sciences Centre ( Site 2806), London, Ontario
  - The Ottawa Hospital - General Campus ( Site 2813), Ottawa, Ontario
  - Sunnybrook Research Institute ( Site 2802), Toronto, Ontario
  - Mount Sinai Hospital ( Site 2811), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 2803), Toronto, Ontario
  - Centre Intégré de Santé et de Services Sociaux de la Montérégie-Centre-Oncology ( Site 2809), Greenfield Park, Quebec
  - Centre Intégré de Santé et de Services Sociaux (CISSS) de La-Centre intégré de cancérologie de Lava ( Site 2810), Laval, Quebec
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 2807), Montreal, Quebec
  - Jewish General Hospital ( Site 2800), Montreal, Quebec
  - St. Marys Hospital Center ( Site 2820), Montreal, Quebec
  - McGill University Health Centre ( Site 2818), Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 2805), Québec, Quebec
  - Centre intégré universitaire de santé et de services sociaux de l'Estrie - Centre Hospitalier Univer ( Site 2812), Sherbrooke, Quebec
  - Centre integre universitaire de sante et de services sociaux de la Mauricie-et-du-centre-du-quebec ( Site 2816), Trois-Rivières, Quebec
- Chile (16):
  - IC La Serena Research ( Site 2766), La Serena, Coquimbo Region
  - UNIVERSIDAD CATÓLICA DEL MAULE ( Site 2768), Talca, Maule Region
  - Centro de Estudios Clínicos SAGA ( Site 2767), Santiago, Region M. de Santiago
  - Orlandi Oncologia-Oncology ( Site 2752), Santiago, Region M. de Santiago
  - Fundacion Arturo Lopez Perez FALP ( Site 2750), Santiago, Region M. de Santiago
  - Oncovida ( Site 2759), Santiago, Region M. de Santiago
  - Clínica Inmunocel ( Site 2762), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile-Hemato-Oncology ( Site 2751), Santiago, Region M. de Santiago
  - Instituto Nacional del Cancer-CR Investigación ( Site 2753), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 2756), Santiago, Region M. de Santiago
  - James Lind Centro de Investigacion del Cancer ( Site 2757), Temuco, Región de la Araucanía
  - CIDO SpA ( Site 2765), Temuco, Región de la Araucanía
  - ONCOCENTRO APYS-ACEREY ( Site 2758), Viña del Mar, Región de Valparaíso
  - Centro de Investigaciones ( Site 2755), Viña del Mar, Región de Valparaíso
  - Biocenter ( Site 2763), Concepción, Región del Biobío
  - Bradford Hill Norte ( Site 2761), Antofagasta
- China (56):
  - Anhui Provincial Hospital-Cancer Chemotherapy Department ( Site 3480), Hefei, Anhui
  - Anhui Provincil Hospital South District-Respiratory Medicine Dept ( Site 3487), Hefei, Anhui
  - Beijing Cancer Hospital ( Site 3451), Beijing, Beijing Municipality
  - The Fifth Medical Center Of The Chinese PLA General Hospital (South) ( Site 3465), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 3499), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 3500), Beijing, Beijing Municipality
  - Beijing Cancer hospital-Thoracic Cancer Department A ( Site 3454), Beijing, Beijing Municipality
  - Chinese Academy of medical science, Peking Union Medical College Hospital(Dongdan) ( Site 3466), Beijing, Beijing Municipality
  - Army Medical Center of People's Liberation Army-Oncology Department ( Site 3477), Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital ( Site 3461), Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University ( Site 3514), Xiamen, Fujian
  - Southern medical university Nangfang Hospital ( Site 3490), Guanghzou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University ( Site 3491), Guangzhou, Guangdong
  - SUN YAT-SEN UNIVERSITY CANCER CENTRE-Internal Medicine ( Site 3452), Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center-melanoma ( Site 3482), Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital-Cancer Center ( Site 3462), Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University-pneumology department ( Site 3459), Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University-thoracic surgery department ( Site 3460), Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University ( Site 3509), Guangzhou, Guangdong
  - The Affiliated Cancer Hospital of Guizhou Medical University ( Site 3498), Guiyang, Guizhou
  - Harbin Medical University Cancer Hospital ( Site 3506), Harbin, Heilongjiang
  - Harbin Medical University Cancer Hospital-Harbin Medical University Cancer Hospital ( Site 3475), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 3488), Zhengzhou, Henan
  - Tongji Hospital Tongji Medical,Science & Technology-oncology ( Site 3476), Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology ( Site 3492), Wuhan, Hubei
  - Xiangya Hospital Central South University ( Site 3508), Changsha, Hunan
  - Xiangya Hospital Central South University-Gynecology ( Site 3497), Changsha, Hunan
  - Xiangya Hospital Central South University-Respiratory ( Site 3479), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 3485), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 3501), Changsha, Hunan
  - Jiangsu Cancer Hospital-Medical Oncotherapy ( Site 3469), Nanjing, Jiangsu
  - Yancheng First People s Hospital ( Site 3504), Yancheng, Jiangsu
  - Northern Jiangsu People's Hospital-General Surgery Department ( Site 3474), Yangzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University ( Site 3513), Nanchang, Jiangxi
  - The First Hospital of Jilin University-Oncology ( Site 3464), Changchun, Jilin
  - Jilin Province Tumor Hospital ( Site 3484), Changchun, Jilin
  - Tangdu Hospital of Fourth Military Medical University of Chi-department of radiotherapy ( Site 3455), Xi'an, Shaanxi
  - Shandong Cancer Hospital ( Site 3517), Jinan, Shandong
  - LinYi Cancer Hospital ( Site 3511), Linyi, Shandong
  - Fudan University Shanghai Cancer Center ( Site 3467), Shanghai, Shanghai Municipality
  - Zhongshan Hospital of Fudan University ( Site 3503), Shanghai, Shanghai Municipality
  - Obstetrics & Gynecology Hospital of Fudan University ( Site 3494), Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital ( Site 3470), Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi an Jiaotong University ( Site 3489), XiAn, Shanxi
  - West China Hospital Sichuan University-respiratory ( Site 3473), Chengdu, Sichuan
  - Sichuan Cancer hospital. ( Site 3515), Chengdu, Sichuan
  - The Second People's Hospital of Yibin ( Site 3516), Yibin, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital ( Site 3456), Tianjin, Tianjin Municipality
  - Xinjiang Medical University Cancer Hospital - Urumqi-galactophore department ( Site 3486), Ürümqi, Xinjiang
  - The Affiliated Cancer Hospital of Xinjiang Medical University ( Site 3502), Ürümqi, Xinjiang
  - Women s Hospital School of Medicine Zhejiang University ( Site 3493), Hangzhou, Zhejiang
  - Hangzhou Cancer Hospital-Medical Oncology ( Site 3468), Hangzhou, Zhejiang
  - The First Affiliated Hospital of Zhejiang University ( Site 3518), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 3495), Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital ( Site 3505), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 3481), Hangzhou, Zhejiang
- Colombia (10):
  - Instituto de Cancerología-Oncology ( Site 2702), Medellín, Antioquia
  - Fundacion Colombiana de Cancerología Clinica Vida ( Site 2707), Medellín, Antioquia
  - Clinica de la Costa S.A.S. ( Site 2705), Barranquilla, Atlántico
  - Administradora Country S.A. ( Site 2701), Bogotá, Bogota D.C.
  - Sociedad De Oncología y Hematología Del Cesar SAS-Oncology ( Site 2704), Valledupar, Cesar Department
  - Instituto Nacional De Cancerologia-Oncología Clínica ( Site 2706), Bogota, Cundinamarca
  - IMAT S.A.S ( Site 2703), Montería, Departamento de Córdoba
  - Oncologos del Occidente ( Site 2709), Pereira, Risaralda Department
  - Fundación Valle del Lili ( Site 2700), Cali, Valle del Cauca Department
  - Clínica Imbanaco S.A.S ( Site 2708), Cali, Valle del Cauca Department
- Costa Rica (2):
  - Hospital Metropolitano - Sede Lindora ( Site 3901), Santa Ana, Provincia de San José
  - CIMCA ( Site 3900), San José
- Czechia (6):
  - Masarykuv onkologicky ustav-Klinika komplexni onkologicke pece ( Site 0703), Brno, Brno-mesto
  - Fakultni nemocnice Olomouc-Onkologicka klinika ( Site 0704), Olomouc, Olomoucký kraj
  - Fakultni Thomayerova nemocnice-Onkologicka klinika 1. LF UK ( Site 0702), Prague, Praha 4
  - Fakultni nemocnice v Motole-Onkologicka klinika 2. LF UK a FN Motol ( Site 0705), Prague, Praha 5
  - Fakultni nemocnice Olomouc ( Site 0701), Olomouc
  - Fakultni nemocnice v Motole ( Site 0700), Prague
- Denmark (2):
  - Odense Universitetshospital ( Site 0650), Odense, Region Syddanmark
  - Vejle Sygehus ( Site 0653), Vejle, Region Syddanmark
- Tartu University Hospital-Radiotherapy and oncology ( Site 3800), Tartu, Tartu, Estonia
- Finland (2):
  - Tampere University Hospital [Tampere Finland] ( Site 0600), Tampere, Pirkanmaa
  - Turku University Hospital ( Site 0601), Turku, Southwest Finland
- France (49):
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet-Dermatology Department ( Site 2539), Nice, Alpes-Maritimes
  - Nouvel Hôpital Civil (NHC) ( Site 2529), Strasbourg, Alsace
  - CHU Bordeaux Haut-Leveque ( Site 2534), Pessac, Aquitaine
  - CH Lyon Sud Hospices Civils de Lyon ( Site 2521), Pierre-Bénite, Auvergne-Rhône-Alpes
  - Centre Hopitalar Leon-Berard ( Site 2519), Lyon, Auvergne
  - Hopital Nord ( Site 2516), Marseille, Bouches-du-Rhone
  - Hôpital Privé Clairval ( Site 2549), Marseille, Bouches-du-Rhone
  - CHU La Timone ( Site 2508), Marseille, Bouches-du-Rhone
  - Centre Francois Baclesse ( Site 2558), Caen, Calvados
  - Centre Georges François Leclerc-Centre de recherche clinique ( Site 2536), Dijon, Cote-d Or
  - CHU-Jean Minjoz ( Site 2550), Besançon, Doubs
  - CHU Jean Minjoz ( Site 2520), Besançon, Doubs
  - CHRU Brest - Hopital Cavale Blanche ( Site 2504), Brest, Finistere
  - Institut Bergonie ( Site 2502), Bordeaux, Gironde
  - CHU Toulouse - Hopital Rangueil ( Site 2518), Toulouse, Haute-Garonne
  - Institut Universitaire du Cancer Toulouse - Oncopole - CHU de TOULOUSE ( Site 2560), Toulouse, Haute-Garonne
  - CHU de Toulouse - Hopital Larrey-service de pneumologie ( Site 2526), Toulouse, Haute-Garonne
  - Centre Hospitalier Annecy Genevois ( Site 2554), Epagny Metz Tessy, Haute-Savoie
  - Centre Oscar Lambret ( Site 2551), Lille, Hauts-de-France
  - Ambroise Pare Hopital ( Site 2503), Boulogne, Hauts-de-Seine
  - Hôpital Foch ( Site 2543), Suresnes, Hauts-de-Seine
  - CHU Montpellier. ( Site 2556), Montpellier, Herault
  - Centre Eugène Marquis Rennes - Centre de Lutte Contre le Cancer ( Site 2525), Rennes, Ille-et-Vilaine
  - Hopital Trousseau ( Site 2512), Chambray-lès-Tours, Indre-et-Loire
  - C.H.U. de Tours - Hopital Bretonneau ( Site 2515), Tours, Indre-et-Loire
  - Hôpital Nord Guillaume-et-René-Laennec / CHU de Nantes-lung oncology ( Site 2546), Saint-Herblain, Loire-Atlantique
  - Institut de Cancérologie de l'Ouest-Oncologie Médicale ( Site 2522), Saint-Herblain, Loire-Atlantique
  - Institut de Cancérologie de Lorraine Alexis Vautrin ( Site 2532), Vandœuvre-lès-Nancy, Lorraine
  - CHRU Lille Hospital Claude Huriez ( Site 2506), Lille, Nord
  - Centre Jean Perrin - Centre Régional de Lutte contre le Cancer d'Auvergne-ONCOLOGY ( Site 2542), Clermont-Ferrand, Puy-de-Dome
  - Centre Hospitalier de Pau ( Site 2563), Pau, Pyrenees-Atlantiques
  - C.H.U. Pontchaillou ( Site 2511), Pierre-Bénite, Rhone
  - Centre Hospitalier du Mans-Pneumologie ( Site 2527), Le Mans, Sarthe
  - Centre Henri Becquerel ( Site 2547), Rouen, Seine-Maritime
  - Hôpital Avicenne-Dermatologie ( Site 2538), Bobigny, Seine-Saint-Denis
  - Clinique de L'Europe ( Site 2548), Amiens, Somme
  - Centre Hopitalier Intercommunal Creteil ( Site 2514), Créteil, Val-de-Marne
  - HENRI MONDOR HOSPITAL ( Site 2561), Créteil, Val-de-Marne
  - Hôpital Universitaire Paul Brousse ( Site 2541), Villejuif, Val-de-Marne
  - Institut Sainte Catherine ( Site 2557), Avignon, Vaucluse
  - Centre Hospitalier Universitaire de Poitiers-Dermatologie ( Site 2544), Poitiers, Vienne
  - Hopital Cochin ( Site 2509), Paris
  - Hopital Saint Louis ( Site 2510), Paris
  - CHU Hopital Saint Antoine ( Site 2517), Paris
  - Groupe Hospitalier Diaconesses Croix Saint Simon ( Site 2545), Paris
  - Hôpital Tenon ( Site 2530), Paris
  - Hôpital Beaujon ( Site 2524), Clichy, Île-de-France Region
  - Groupe hospitalier Paris saint Joseph-Service de Pneumologie-Allergologie -Oncologie Thoracique ( Site 2533), Paris, Île-de-France Region
  - Institut Gustave Roussy ( Site 2513), Villejuif, Île-de-France Region
- Germany (13):
  - Universitaetsklinikum Tuebingen ( Site 2405), Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Erlangen ( Site 2408), Erlangen, Bavaria
  - Universitaetsklinik Muenchen ( Site 2406), Munich, Bavaria
  - Krankenhaus Nordwest ( Site 2409), Frankfurt am Main, Hesse
  - Elbe Klinikum Buxtehude ( Site 2400), Buxtehude, Lower Saxony
  - Medizinische Hochschule Hannover ( Site 2402), Hanover, Lower Saxony
  - Universitaetsklinikum Essen ( Site 2404), Essen, North Rhine-Westphalia
  - Universitaetsklinikum des Saarlandes-Klinik für Innere Medizin V-Pneumologie, Allergologie, Beatmun ( Site 2411), Homburg, Saarland
  - Universitatsklinikum Carl Gustav Carus ( Site 2407), Dresden, Saxony
  - LungenClinic Grosshansdorf GmbH ( Site 2412), Großhansdorf, Schleswig-Holstein
  - SRH Wald-Klinikum Gera GmbH ( Site 2403), Gera, Thuringia
  - Helios Klinikum Emil von Behring Berlin-Zehlendorf-Lungenklinik Heckeshorn ( Site 2418), Berlin
  - Facharztzentrum Eppendorf ( Site 2415), Hamburg
- Greece (4):
  - General Hospital of Athens "Laiko"-Hematology Department ( Site 1851), Athens, Attica
  - Sotiria Regional Chest Diseases Hospital of Athens ( Site 1850), Athens, Attica
  - Andreas Syggros Hospital ( Site 1853), Athens, Attica
  - European Interbalkan Medical Center ( Site 1855), Thessaloniki
- Guatemala (4):
  - MEDI-K ( Site 3403), Guatemala City
  - CELAN,S.A ( Site 3405), Guatemala City
  - Oncomedica ( Site 3401), Guatemala City
  - Grupo Medico Angeles ( Site 3402), Guatemala City
- Hong Kong (3):
  - Queen Mary Hospital ( Site 1902), Hksar
  - Queen Mary Hospital-Department of Medicine (Respiratory) ( Site 1900), Hksar
  - Princess Margaret Hospital ( Site 1903), Hong Kong
- Hungary (18):
  - Békés Megyei Központi Kórház Pándy Kálmán Tagkórház-Megyei Onkológiai Centrum ( Site 1405), Gyula, Bekes County
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Oktatókórház ( Site 1409), Miskolc, Borsod-Abauj Zemplen county
  - Bacs-Kiskun Varmegyei Oktatokorhaz-Onkoradiologiai Kozpont ( Site 1419), Kecskemét, Bács-Kiskun county
  - Fejér Megyei Szent György Egyetemi Oktató Kórház-l.Pulmonologia ( Site 1407), Székesfehérvár, Fejér
  - Petz Aladar Egyetemi Oktato Korhaz-Pulmonológia (Dr. Szalai Zsuzsanna) ( Site 1408), Győr, Győr-Moson-Sopron
  - Mátrai Gyógyintézet ( Site 1417), Gyöngyös, Heves County
  - Jász-Nagykun-Szolnok Vármegyei Hetényi Géza Kórház ( Site 1401), Szolnok, Jász-Nagykun-Szolnok
  - Országos Onkológiai Intézet-Urogenitális Tumorok és Klinikai Farmakológiai Osztály ( Site 1411), Budapest, Pest County
  - Reformatus Pulmonologiai Centrum ( Site 1418), Törökbálint, Pest County
  - Markusovszky Egyetemi Oktatokorhaz-Onkológiai Osztály ( Site 1410), Szombathely, Vas County
  - Farkasgyepui Tudogyogyintezet-Pulmonologia ( Site 1414), Farkasgyepű, Veszprém megye
  - Semmelweis University-Belgyógyászati és Hematológiai Klinika ( Site 1406), Budapest
  - Orszagos Koranyi Pulmonologiai Intezet ( Site 1403), Budapest
  - Uzsoki Utcai Kórház-Onkoradiológiai Osztály ( Site 1413), Budapest
  - Debreceni Egyetem Klinikai Kozpont-Belgyógyászati Klinika (Haematologia) ( Site 1415), Debrecen
  - Debreceni Egyetem Klinikai Kozpont-Onkológiai Klinika ( Site 1412), Debrecen
  - Somogy Megyei Kaposi Mor Oktato Korhaz ( Site 1402), Kaposvár
  - Zala Megyei Szent Rafael Korhaz ( Site 1400), Zalaegerszeg
- Ireland (3):
  - Mater Misercordiae University Hospital ( Site 1800), Dublin, Leinster
  - Tallaght University Hospital ( Site 1803), Dublin
  - St. James s Hospital ( Site 1801), Dublin
- Israel (12):
  - Rambam Health Care Campus-Oncology Division ( Site 2053), Haifa
  - Bnai Zion Medical Center ( Site 2060), Haifa
  - Shaare Zedek Medical Center ( Site 2068), Jerusalem
  - Hadassah Ein Kerem Medical Center ( Site 2051), Jerusalem
  - Rabin Medical Center ( Site 2059), Petah Tikva
  - Chaim Sheba Medical Center. ( Site 2052), Ramat Gan
  - Chaim Sheba Medical Center ( Site 2055), Ramat Gan
  - Sheba Medical Center ( Site 2062), Ramat Gan
  - Sheba Medical Center ( Site 2065), Ramat Gan
  - ZIV Medical Center-Hematology Institute ( Site 2061), Safed
  - Sourasky Medical Center ( Site 2054), Tel Aviv
  - Shamir Medical Center Assaf Harofeh ( Site 2058), Ẕerifin
- Italy (26):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola ( Site 1978), Bologna, Emilia-Romagna
  - Istittuto Nazionale dei Tumori Regina Elena IRCCS - IFO ( Site 1963), Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS -Medical Oncology ( Site 1975), Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 1977), Milan, Lombardy
  - Azienda Ospedaliera San Gerardo ( Site 1980), Monza, Lombardy
  - Humanitas-U.O di Oncologia medica ed Ematologia ( Site 1968), Rozzano, Milano
  - IRCCS CRO Aviano, Hematology/Oncology ( Site 1957), Aviano, Pordenone
  - Ospedale Cannizzaro ( Site 1981), Catania, Sicily
  - Istituto di Candiolo - IRCCS ( Site 1960), Candiolo, Torino
  - Ospedale San Luigi Gonzaga ( Site 1956), Orbassano, Torino
  - AO Santa Maria della Misericordia-Oncology Department ( Site 1971), Perugia, Umbria
  - Istituto Oncologico Veneto IRCCS ( Site 1976), Padua, Veneto
  - Humanitas Gavazzeni ( Site 1954), Bergamo
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII-UOC Oncologia ( Site 1967), Bergamo
  - Azienda Ospedaliera Spedali Civili di Brescia-Oncology ( Site 1972), Brescia
  - IRCCS A.O.U. San Martino - IST ( Site 1961), Genova
  - Ospedale San Raffaele. ( Site 1979), Milan
  - Istituto Europeo di Oncologia ( Site 1952), Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 1955), Napoli
  - Azienda Ospedaliero Universitaria di Parma-UO Oncologia Medica ( Site 1964), Parma
  - Fondazione IRCCS Policlinico San Matteo ( Site 1982), Pavia
  - Azienda Ospedaliera San Camillo Forlanini ( Site 1958), Roma
  - Policlinico Universitario Agostino Gemelli ( Site 1965), Roma
  - ospedale le scotte-U.O.C. Immunoterapia Oncologica ( Site 1969), Siena
  - Azienda Ospedaliera Santa Maria ( Site 1962), Terni
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino ( Site 1974), Torino
- Japan (85):
  - National Hospital Organization Nagoya Medical Center ( Site 3109), Nagoya, Aichi-ken
  - Aichi Cancer Center ( Site 3101), Nagoya, Aichi-ken
  - Nagoya University Hospital ( Site 3151), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 3121), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 3116), Matsuyama, Ehime
  - Ehime University Hospital ( Site 3158), Tōon, Ehime
  - Kurume University Hospital ( Site 3105), Kurume, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center ( Site 3160), Sapporo, Hokkaido
  - Sapporo Kosei General Hospital ( Site 3172), Sapporo, Hokkaido
  - Sapporo Medical University Hospital ( Site 3113), Sapporo, Hokkaido
  - Hokkaido University Hospital ( Site 3165), Sapporo, Hokkaido
  - Hyogo Cancer Center ( Site 3131), Akashi, Hyōgo
  - National Hospital Organization Himeji Medical Center ( Site 3111), Himeji, Hyōgo
  - Kobe City Medical Center General Hospital ( Site 3144), Kobe, Hyōgo
  - Hyogo Medical University Hospital ( Site 3100), Nishinomiya, Hyōgo
  - Ibaraki Prefectural Central Hospital ( Site 3180), Kasama, Ibaraki
  - University of Tsukuba Hospital ( Site 3176), Tsukuba, Ibaraki
  - Kanazawa University Hospital ( Site 3140), Kanazawa, Ishikawa-ken
  - Iwate Medical University Hospital ( Site 3157), Shiwa-gun, Iwate
  - Kagawa University Hospital ( Site 3171), Kita, Kagawa-ken
  - Nippon Medical School Musashi Kosugi Hospital ( Site 3178), Kawasaki, Kanagawa
  - St. Marianna University Hospital ( Site 3182), Kawasaki, Kanagawa
  - Kitasato University Hospital ( Site 3142), Sagamihara, Kanagawa
  - Yokohama City University Hospital ( Site 3163), Yokohama, Kanagawa
  - Kanagawa Cancer Center ( Site 3137), Yokohama, Kanagawa
  - Yokosuka Kyosai Hospital ( Site 3150), Yokosuka, Kanagawa
  - Miyagi Cancer Center ( Site 3122), Natori-shi, Miyagi
  - Tohoku University Hospital ( Site 3175), Sendai, Miyagi
  - Sendai Kousei Hospital ( Site 3115), Sendai, Miyagi
  - Nara Medical University Hospital ( Site 3110), Kashihara, Nara
  - Niigata Cancer Center Hospital ( Site 3173), Niigata, Niigata
  - Kurashiki Central Hospital ( Site 3132), Kurashiki, Okayama-ken
  - University of the Ryukyus Hospital ( Site 3155), Ginowan, Okinawa
  - Osaka Habikino Medical Center ( Site 3138), Habikino, Osaka
  - Kansai Medical University Hospital ( Site 3126), Hirakata, Osaka
  - Kindai University Hospital ( Site 3102), Sakai, Osaka
  - Kindai University Hospital ( Site 3135), Sakai, Osaka
  - Kindai University Hospital ( Site 3166), Sakai, Osaka
  - Osaka Rosai Hospital ( Site 3148), Sakai, Osaka
  - The University of Osaka Hospital ( Site 3168), Suita, Osaka
  - Osaka Medical and Pharmaceutical University Hospital ( Site 3167), Takatsuki, Osaka
  - Osaka Medical and Pharmaceutical University Hospital ( Site 3187), Takatsuki, Osaka
  - Saitama Medical University International Medical Center ( Site 3118), Hidaka, Saitama
  - Saitama Prefectural Cancer Center ( Site 3112), Kitaadachi-gun, Saitama
  - Dokkyo Medical University Saitama Medical Center ( Site 3152), Koshigaya, Saitama
  - National Defense Medical College Hospital ( Site 3177), Tokorozawa, Saitama
  - Shizuoka Cancer Center ( Site 3128), Nakatogari, Shizuoka
  - Jichi Medical University Hospital ( Site 3141), Shimotsuke, Tochigi
  - Institute of Science Tokyo Hospital ( Site 3149), Bunkyō, Tokyo
  - Cancer Institute Hospital of JFCR ( Site 3146), Koto, Tokyo
  - Cancer Institute Hospital of JFCR ( Site 3164), Koto, Tokyo
  - Toranomon Hospital ( Site 3134), Minato-ku, Tokyo
  - Toranomon Hospital ( Site 3153), Minato-ku, Tokyo
  - Kyorin University Hospital ( Site 3103), Mitaka, Tokyo
  - Kyorin University Hospital ( Site 3147), Mitaka-shi, Tokyo
  - Tokyo Medical University Hospital ( Site 3170), Shinjuku-ku, Tokyo
  - National Hospital Organization Yamaguchi Ube Medical Center ( Site 3123), Ube, Yamaguchi
  - Yamaguchi University Hospital ( Site 3114), Ube, Yamaguchi
  - Chiba Cancer Center ( Site 3117), Chiba
  - National Hospital Organization Kyushu Medical Center ( Site 3136), Fukuoka
  - National Hospital Organization Kyushu Cancer Center ( Site 3169), Fukuoka
  - Kyushu University Hospital ( Site 3143), Fukuoka
  - Kyushu University Hospital ( Site 3185), Fukuoka
  - Gifu University Hospital ( Site 3161), Gifu
  - Hiroshima City Hiroshima Citizens Hospital ( Site 3119), Hiroshima
  - Hiroshima University Hospital ( Site 3154), Hiroshima
  - Kochi Health Sciences Center ( Site 3145), Kochi
  - Kumamoto University Hospital ( Site 3179), Kumamoto
  - Kyoto University Hospital ( Site 3181), Kyoto
  - Niigata University Medical & Dental Hospital ( Site 3174), Niigata
  - Okayama University Hospital ( Site 3107), Okayama
  - Osaka City General Hospital ( Site 3125), Osaka
  - National Hospital Organization Osaka National Hospital ( Site 3162), Osaka
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute ( Site 3129), Osaka
  - Osaka General Medical Center ( Site 3184), Osaka
  - National Cancer Center Hospital ( Site 3130), Tokyo
  - St.Luke's International Hospital ( Site 3120), Tokyo
  - The Jikei University Hospital ( Site 3156), Tokyo
  - Nippon Medical School Hospital ( Site 3139), Tokyo
  - Tokyo Metropolitan Komagome Hospital ( Site 3133), Tokyo
  - Cancer Institute Hospital of JFCR ( Site 3108), Tokyo
  - Keio University Hospital ( Site 3127), Tokyo
  - Teikyo University Hospital ( Site 3104), Tokyo
  - Toyama Prefectural Central Hospital ( Site 3183), Toyama
  - Wakayama Medical University Hospital ( Site 3124), Wakayama
- Latvia (2):
  - Liepjas reionl slimnca ( Site 3851), Liepāja
  - RIGA EAST UNIVERSITY HOSPITAL ,Oncology Centre of Latvia-Out-patient and Day patient facility of Ch ( Site 3850), Riga
- Lithuania (3):
  - Klaipeda University Hospital-Oncology chemotherapy ( Site 3302), Klaipėda, Klaipedos Miestas
  - Vilniaus Universiteto Ligonine Santaros Klinikos ( Site 3300), Vilnius
  - Vilnius University Hospital Santaros Clinics Affiliate - National Cancer Center ( Site 3301), Vilnius
- Malaysia (6):
  - Hospital Tengku Ampuan Afzan ( Site 0627), Kuantan, Pahang
  - Gleneagles Penang ( Site 0625), George Town, Pulau Pinang
  - Hospital Pulau Pinang ( Site 0629), George Town, Pulau Pinang
  - Institut Kanser Negara - National Cancer Institute ( Site 0630), Putrajaya - Wilayah Persekutuan, Putrajaya
  - Pantai Hospital Kuala Lumpur ( Site 0628), Kuala Lumpur
  - University Malaya Medical Centre ( Site 0626), Kuala Lumpur
- Mexico (14):
  - Investigación Oncofarmacéutica-Investigación clínica ( Site 1114), La Paz, Baja California Sur
  - Centro de Inmuno Oncología de Occidente SA de CV ( Site 1115), Guadalajara, Jalisco
  - Arke Estudios Clinicos ( Site 1117), Mexico City, Mexico City
  - INSTITUTO NACIONAL DE CANCEROLOGIA ( Site 1102), Mexico City, Mexico City
  - Avix Investigación Clinica, S.C.-Oncology ( Site 1104), Monterrey, Nuevo León
  - I Can Oncology Center SA de CV ( Site 1116), Monterrey, Nuevo León
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez"-Hematologia and Oncologia ( Site 1113), Monterrey, Nuevo León
  - Centro de Urologa Avanzada del Noreste ( Site 1110), San Pedro Garza García, Nuevo León
  - Oaxaca Site Management Organization ( Site 1106), Oaxaca City, Oaxaca
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, S.C. ( Site 1119), Ciudad Madero, Tamaulipas
  - Medical Care and Research SA de CV ( Site 1103), Mérida, Yucatán
  - Unidad de Mastologia Avanzada de Chihuahua S.A de C.V ( Site 1109), Chihuahua City
  - Oncare Viaducto Napoles ( Site 1107), Mexico City
  - Cuidados Oncologicos. ( Site 1118), Querétaro
- Netherlands (5):
  - Radboud University Medical Center ( Site 1554), Nijmegen, Gelderland
  - Antoni van Leeuwenhoek Ziekenhuis ( Site 1551), Amsterdam, North Holland
  - Amsterdam UMC, locatie VUmc ( Site 1555), Amsterdam, North Holland
  - Erasmus MC ( Site 1553), Rotterdam, South Holland
  - Universitair Medisch Centrum Groningen ( Site 1550), Groningen
- New Zealand (5):
  - Canterbury Regional Cancer & Blood Service ( Site 1500), Christchurch, Canterbury
  - Palmerston North Hospital, MidCentral DHB ( Site 1504), Palmerston North, Manawatu-Wanganui
  - Waikato Hospital ( Site 1502), Hamilton, Waikato Region
  - Auckland City Hospital ( Site 1503), Auckland
  - Capital & Coast District Health Board - Wellington Hospital ( Site 1501), Wellington
- Norway (3):
  - Helse Bergen Haukeland universitetssykehus ( Site 1451), Bergen, Vestfold
  - Oslo Universitetssykehus Radiumhospitalet ( Site 1450), Oslo
  - Oslo universitetssykehus, Radiumhospitalet ( Site 1452), Oslo
- Peru (3):
  - IPOR Instituto Peruano de Oncología & Radioterapia ( Site 0678), Lima
  - INSTITUTO NACIONAL DE ENFERMEDADES NEOPLASICAS ( Site 0681), Lima
  - Hospital Cayetano Heredia-Oncology ( Site 0675), Lima
- Philippines (3):
  - Makati Medical Center ( Site 1702), Makati City, National Capital Region
  - Lung Center of the Philippines ( Site 1705), Quezon City, National Capital Region
  - St. Luke s Medical Center ( Site 1700), Quezon City, National Capital Region
- Poland (21):
  - Przychodnia Lekarska KOMED ( Site 1603), Konin, Greater Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny w Poznaniu ( Site 1607), Poznan, Greater Poland Voivodeship
  - Med-Polonia Sp. z o. o. ( Site 1605), Poznan, Greater Poland Voivodeship
  - Szpital Kliniczny im. Przemienienia Panskiego Uniwersytetu Medycznego im. K. Marcinkowskiego w Pozna ( Site 1601), Poznan, Greater Poland Voivodeship
  - Wielkopolskie Centrum Onkologii im.M.Sklodowskiej-Curie ( Site 1619), Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 1612), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Oddzial w Krakowie ( Site 1608), Krakow, Lesser Poland Voivodeship
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie-Oncology Department ( Site 1618), Krakow, Lesser Poland Voivodeship
  - Luxmed Onkologia sp. z o. o. ( Site 1621), Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie ( Site 1604), Warsaw, Masovian Voivodeship
  - Wojskowy Instytut Medyczny-Klinika Onkologii ( Site 1606), Warsaw, Masovian Voivodeship
  - Opolskie Centrum Onkologii w Opolu im. prof. Tadeusza Kosza-Klinika Onkologii z Odcinkiem Dziennym ( Site 1616), Opole, Opole Voivodeship
  - Bialostockie Centrum Onkologii ( Site 1610), Bialystok, Podlaskie Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Klinika Chirurgii Onkologicznej, Transplantacyjnej i Ogólnej ( Site 1622), Gdansk, Pomeranian Voivodeship
  - Szpital Morski im. PCK. Szpitale Pomorskie Sp. Z o.o ( Site 1625), Gdynia, Pomeranian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach ( Site 1620), Gliwice, Silesian Voivodeship
  - Szpital Rejonowy im. dr. J. Rostka w Raciborzu ( Site 1624), Racibórz, Silesian Voivodeship
  - Warminsko-Mazurskie Centrum Chorob Pluc w Olsztynie ( Site 1623), Olsztyn, Warmian-Masurian Voivodeship
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie ( Site 1614), Koszalin, West Pomeranian Voivodeship
  - Powiatowe Centrum Zdrowia w Brzezinach Sp. z o. o. Oddział Dziennej Chemioterapii ( Site 1611), Brzeziny, Łódź Voivodeship
  - Instytut Centrum Zdrowia Matki Polki-Klinika Onkologii ( Site 1609), Lodz, Łódź Voivodeship
- Portugal (4):
  - Champalimaud Foundation ( Site 1751), Lisbon, Lisbon District
  - Unidade Local de Saude de Santa Maria - Hospital Pulido Valente ( Site 1750), Lisbon
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE-Oncologia Médica ( Site 1753), Porto
  - Centro Hospitalar de Sao Joao - Hospital de Sao Joao ( Site 1752), Porto
- Puerto Rico (3):
  - Ad-Vance Medical Research-Research ( Site 1151), Ponce
  - FDI Clinical Research ( Site 1152), San Juan
  - UPR Comprehensive Cancer Center ( Site 1150), San Juan
- Romania (6):
  - MEMORIAL HEALTHCARE INTERNATIONAL S.R.L ( Site 3553), Bucharest, București
  - Cardiomed SRL Cluj-Napoca ( Site 3555), Cluj-Napoca, Cluj
  - Centrul de Oncologie "Sfântul Nectarie" ( Site 3552), Craiova, Dolj
  - Cabinet Medical Oncomed ( Site 3554), Timișoara, Timiș County
  - Institutul Oncologic "Prof. Dr. Ioan Chiricuta" ( Site 3551), Cluj-Napoca
  - Spitalul Județean Sfântul Ioan cel Nou Suceava-Oncology ( Site 3550), Suceava
- Russia (37):
  - Altai Regional Clinical Oncology Center ( Site 1229), Barnaul, Altayskiy Kray
  - GBUZ Republican Clinical Oncological Dispensary-Antitumor drug therapy department ( Site 1250), Ufa, Baskortostan, Respublika
  - Republican Clinical Oncology Dispensary of Republic of Bashkortostan ( Site 1204), Ufa, Baskortostan, Respublika
  - Bashkir State Medical University ( Site 1221), Ufa, Baskortostan, Respublika
  - Belgorod Oncology Dispensary ( Site 1213), Belgorod, Belgorod Oblast
  - LLC Medical Centre "Lotos" ( Site 1253), Chelyabinsk, Chelyabinsk Oblast
  - Regional Budgetary Healthcare Institution 'Ivanovo Regional Oncology Dispensary'-Urology ( Site 1219), Ivanovo, Ivanovo Oblast
  - Oncological Dispensary #2 of Ministry of Health of Krasnodar region ( Site 1244), Sochi, Krasnodarskiy Kray
  - GBUZ LOKB ( Site 1218), Saint-Petersburg, Leningradskaya Oblast'
  - GBUZ LOKB-Oncology department #1 ( Site 1222), Saint-Petersburg, Leningradskaya Oblast'
  - Ogarev Mordovia State University ( Site 1206), Saransk, Mordoviya, Respublika
  - The National Medico-Surgical Center N.I. Pirogov ( Site 1225), Moscow, Moscow
  - N.N. Blokhin NMRCO ( Site 1209), Moscow, Moscow
  - Russian Oncological Research Center n.a. N.N.Blokhin of MoH ( Site 1201), Moscow, Moscow
  - FSBI-FRCC of Special Types Med. Care and Technologies FMBA of Russia ( Site 1234), Moscow, Moscow
  - Russian Scientific Center of Roentgenoradiology ( Site 1215), Moscow, Moscow
  - First Moscow State Medical University n.a. I.M.Sechenov ( Site 1245), Moscow, Moscow
  - P. A. Hertsen Moscow Oncology Research Center ( Site 1214), Moscow, Moscow
  - P. A. Hertsen Moscow Oncology Research Center ( Site 1247), Moscow, Moscow
  - FSAI Treatment and Rehabilitation Centre of the MoH and SD of RF ( Site 1208), Moscow, Moscow
  - Volga District Medical Center Federal Medical and Biological Agency ( Site 1242), Nizhny Novgorod, Nizhny Novgorod Oblast
  - Russian Scientific Research Institute of Hematology and Blood Transfusion-Hematology ( Site 1224), Saint Petersburg, Sankt-Peterburg
  - St. Petersburg Clinical Hospital of Russian Academy Of Sciences ( Site 1235), Saint Petersburg, Sankt-Peterburg
  - EuroCityClinic ( Site 1230), Saint Petersburg, Sankt-Peterburg
  - First Pavlov State Medical University of Saint Petersburg ( Site 1232), Saint Petersburg, Sankt-Peterburg
  - Almazov National Medical Research Centre ( Site 1233), Saint Petersburg, Sankt-Peterburg
  - Clinical Research Center of specialized types medical care-Oncology ( Site 1205), Saint Petersburg, Sankt-Peterburg
  - N.N.Petrov Research Institute of Oncology-Department of Preclinical and Clinical Research ( Site 1211), Saint Petersburg, Sankt-Peterburg
  - National Medical Research Center of Oncology N.A. N.N. Petrov ( Site 1210), Saint Petersburg, Sankt-Peterburg
  - City Clinical Oncology Center ( Site 1237), Saint Petersburg, Sankt-Peterburg
  - GBUZ SK Pyatigorsk Interdistrict Oncology dispensary ( Site 1223), Pyatigorsk, Stavropol Kray
  - Republican Clinical Oncology Dispensary ( Site 1228), Kazan', Tatarstan, Respublika
  - Republican Clinical Oncology Dispensary of Tatarstan MoH named after professor M.Z. Sigal ( Site 1203), Kazan', Tatarstan, Respublika
  - Tomsk Scientific Research Institute of Oncology ( Site 1227), Tomsk, Tomsk Oblast
  - SAIH of the Tyumen region, Multidisciplinary Clinical Medical Center "Medical town" ( Site 1220), Tyumen, Tyumen Oblast
  - Udmurtian Republican Clinical Oncology Center ( Site 1212), Izhevsk, Udmurtiya Republic
  - Yaroslavl Regional SBIH Clinical Oncology Hospital ( Site 1243), Yaroslavl, Yaroslavl Oblast
- Singapore (2):
  - National Cancer Centre Singapore ( Site 2200), Singapore, Central Singapore
  - National University Hospital-Haematology -Oncology Research Group ( Site 2201), Singapore, South West
- South Africa (7):
  - WCR Office ( Site 2002), Johannesburg, Gauteng
  - Wilgers Oncology Centre ( Site 2006), Pretoria, Gauteng
  - LIFE GROENKLOOF-Mary Potter Cancer Centre ( Site 2005), Pretoria, Gauteng
  - Sandton Oncology Medical Group (Pty) Ltd-Research ( Site 2004), Sandton, Gauteng
  - The Oncology Centre ( Site 2000), Durban, KwaZulu-Natal
  - Cape Town Oncology Trials ( Site 2007), Cape Town, Western Cape
  - GVI Oncology ( Site 2008), George, Western Cape
- South Korea (21):
  - Gachon University Gil Medical Center ( Site 0967), Inceon, Incheon
  - Chonnam National University Hwasun Hospital-Hemato-Oncology ( Site 0959), Hwasun, Jeonranamdo
  - National Cancer Center ( Site 0955), Goyang-si, Kyonggi-do
  - CHA Bundang Medical Center CHA University ( Site 0957), Seongnam-si, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 0951), Seongnam-si, Kyonggi-do
  - The Catholic University Of Korea St. Vincent's Hospital ( Site 0968), Suwon, Kyonggi-do
  - Ajou University Hospital ( Site 0969), Suwon, Kyonggi-do
  - Chungbuk National University Hospital ( Site 0961), Cheongju-si, North Chungcheong
  - Gangnam Severance Hospital, Yonsei University Health System ( Site 0966), Gangnam-gu, Seoul
  - Asan Medical Center ( Site 0952), Songpagu, Seoul
  - Keimyung University Dongsan Hospital CRC room 1 ( Site 0960), Daegu, Taegu-Kwangyokshi
  - Kyungpook National University Chilgok Hospital ( Site 0964), Deagu, Taegu-Kwangyokshi
  - Chungnam national university hospital-Department of Internal Medicine ( Site 0958), Daejeon, Taejon-Kwangyokshi
  - Korea University Anam Hospital ( Site 0956), Seoul
  - Seoul National University Hospital ( Site 0953), Seoul
  - Severance Hospital ( Site 0954), Seoul
  - Severance Hospital, Yonsei University Health System ( Site 0962), Seoul
  - Samsung Medical Center ( Site 0950), Seoul
  - Samsung Medical Center ( Site 0970), Seoul
  - Samsung Medical Center ( Site 0971), Seoul
  - Korea University Guro Hospital ( Site 0963), Seoul
- Spain (38):
  - Hospital Universitario Virgen de la Victoria ( Site 0878), Málaga, Andalusia
  - Hospital Universitari Son Espases-Oncologia ( Site 0883), Palma, Balearic Islands
  - Hospital Son Llatzer ( Site 0886), Palma de Mallorca, Balearic Islands
  - Instituto Catalan de Oncologia ICO - Hospital Duran i Reynals ( Site 0860), L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Donostia ( Site 0890), San Sebastian- Donostia, Basque Country
  - H. Marques de Valdecilla ( Site 0865), Santander, Cantabria
  - Institut Catala d Oncologia Hospital Germans Trias i Pujol ( Site 0851), Badalona, Catalonia
  - Hospital Clinic de Barcelona ( Site 0852), Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau-Oncología Médica ( Site 0862), Barcelona, Catalonia
  - CHUS - Hospital Clinico Universitario-Servicio de Oncologia ( Site 0876), Santiago de Compostela, La Coruna
  - Hospital Universitario Insular de Gran Canaria ( Site 0867), Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Puerta de Hierro-Majadahonda ( Site 0861), Majadahonda, Madrid
  - Hospital Universitario Quiron Madrid ( Site 0868), Pozuelo de Alarcón, Madrid
  - Hospital Universitario Ramón y Cajal-Medical Oncology ( Site 0877), Madrid, Madrid, Comunidad de
  - H.R.U Malaga - Hospital General ( Site 0884), Málaga, Malaga
  - Hospital Universitario Central de Asturias-Medical Oncology ( Site 0870), Oviedo, Principality of Asturias
  - Hospital Universitari Sant Joan de Reus-Oncology ( Site 0874), Reus, Tarragona
  - Hospital Universitari i Politecnic La Fe ( Site 0875), Valencia, Valencia
  - Instituto Valenciano de Oncologia - IVO ( Site 0863), Valencia, Valenciana, Comunitat
  - Hospital Clinico de Valencia ( Site 0858), Valencia, Valenciana, Comunitat
  - Hospital General Universitario de Valencia ( Site 0854), Valencia, Valenciana, Comunitat
  - Hospital Arnau de Vilanova ( Site 0866), Valencia, Valenciana, Comunitat
  - Hospital General Universitario de Alicante-Oncologia ( Site 0881), Alicante
  - Parc de Salut Mar - Hospital del Mar-Oncologia ( Site 0873), Barcelona
  - H.U. Vall de Hebron ( Site 0850), Barcelona
  - Hospital Universitario Reina Sofia ( Site 0885), Córdoba
  - Complejo Hospitalario de Jaén-Servicio de Oncología Médica ( Site 0879), Jaén
  - Hospital Universitario Gregorio Maranon ( Site 0864), Madrid
  - Clinica Universitaria de Navarra ( Site 0855), Madrid
  - Hospital Clinico San Carlos ( Site 0857), Madrid
  - Hospital Universitario Fundación Jiménez Díaz-Oncology & Hematology ( Site 0871), Madrid
  - Hospital General Universitario 12 de Octubre ( Site 0856), Madrid
  - Hospital Universitario La Paz ( Site 0853), Madrid
  - Centro Integral Oncologico Clara Campal-Hospital HM Universitario Sanchinarro-START Madrid, ( Site 0869), Madrid
  - Hospital Universitario Virgen Macarena-Unidad de Investigación Oncológica ( Site 0880), Seville
  - HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO-Medical Oncology ( Site 0872), Seville
  - Hospital Universitario Virgen de Valme-Departamento de Oncologia ( Site 0882), Seville
  - Hospital Clinico Universitario Lozano Blesa ( Site 0859), Zaragoza
- Sweden (4):
  - Karolinska Universitetssjukhuset Solna ( Site 0802), Stockholm, Stockholm County
  - Blod och Tumorssjukdomar. Akademiska sjukhuset ( Site 0801), Uppsala, Uppsala County
  - Norrlands Universitetssjukhus ( Site 0800), Umeå, Västerbotten County
  - Sahlgrenska Universitetssjukhuset-Department of Oncology CTU Clinical Trial Unit ( Site 0803), Gothenburg, Västra Götaland County
- Switzerland (3):
  - University Hospital Basel ( Site 0752), Basel, Canton of Basel-City
  - Hôpitaux Universitaires de Genève (HUG) ( Site 0753), Geneva, Canton of Geneva
  - Universitaetsspital Zuerich ( Site 0750), Zürich-Flughafen, Canton of Zurich
- Taiwan (12):
  - Changhua Christian Hospital ( Site 3210), Changhua
  - National Taiwan University Hospital - Hsinchu branch ( Site 3208), Hsinchu
  - Kaohsiung Chang Gung Memorial Hospital ( Site 3203), Kaohsiung City
  - China Medical University Hospital ( Site 3204), Taichung
  - Taichung Veterans General Hospital ( Site 3209), Taichung
  - National Cheng Kung University Hospital ( Site 3201), Tainan
  - National Taiwan University Hospital ( Site 3200), Taipei
  - Mackay Memorial Hospital ( Site 3205), Taipei
  - Taipei Medical University Hospital ( Site 3211), Taipei
  - Taipei Veterans General Hospital ( Site 3202), Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center-Gynecology, Obstetrics, and women's health ( Site 3207), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 3206), Taoyuan District
- Thailand (5):
  - Chulalongkorn University ( Site 2363), Bangkok, Bangkok
  - Ramathibodi Hospital. ( Site 2364), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 2365), Bangkok, Bangkok
  - Faculty of Medicine - Khon Kaen University ( Site 2366), Muang, Changwat Khon Kaen
  - Songklanagarind Hospital ( Site 2367), Hat Yai, Changwat Songkhla
- Turkey (Türkiye) (31):
  - Acibadem Altunizade Hospital-Oncology ( Site 1317), Üsküdar /Istanbul, Istanbul
  - Acibadem Adana Hospital-Pediatric Hematology-Oncology ( Site 1312), Adana
  - Baskent University Dr. Turgut Noyan Research and Training Center-ONCOLOGY ( Site 1307), Adana
  - Adana Sehir Egitim ve Arastirma Hastanesi ( Site 1324), Adana
  - Ankara University Hospital Cebeci ( Site 1306), Ankara
  - Hacettepe Universitesi-oncology hospital ( Site 1304), Ankara
  - Gazi University Health Research and Application Center Gazi Hospital ( Site 1325), Ankara
  - Ankara University Health Practice and Research Hospitals ( Site 1331), Ankara
  - Liv Hospital Ankara ( Site 1330), Ankara
  - Ankara City Hospital-Medical Oncology ( Site 1311), Ankara
  - Baskent Universitesi Ankara Hastanesi ( Site 1303), Ankara
  - Akdeniz Universitesi Hastanesi-Medical Onkology ( Site 1318), Antalya
  - Memorial Antalya Hospital-Oncology ( Site 1315), Antalya
  - Trakya Universitesi Tip Fakultesi ( Site 1301), Edirne
  - Atatürk Üniversitesi ( Site 1333), Erzurum
  - Bezmialem Vakf Üniversitesi-Oncology ( Site 1308), Istanbul
  - Istanbul University Capa Campus ( Site 1314), Istanbul
  - Medipol Mega Universite Hastanesi ( Site 1326), Istanbul
  - Acibadem Universitesi Atakent Hastanesi ( Site 1319), Istanbul
  - Acıbadem Maslak Hastanesi-Medical Oncology ( Site 1321), Istanbul
  - Istanbul Universitesi Cerrahpasa-Medical Oncology ( Site 1302), Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 1316), Istanbul
  - Umraniye Training and Research Hospital ( Site 1329), Istanbul
  - Marmara Universitesi Pendik Egitim Arastirma Hastanesi-Medical Oncology ( Site 1305), Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi ( Site 1300), Izmir
  - Dokuz Eylul Universitesi Hastanesi ( Site 1323), Izmir
  - I.E.U. Medical Point Hastanesi-Oncology ( Site 1310), Izmir
  - Kocaeli Üniversitesi ( Site 1313), Kocaeli
  - Inonu Universitesi ( Site 1309), Malatya
  - Sakarya University School of Medicine ( Site 1332), Sakarya
  - Samsun Medical Park Hastanesi ( Site 1328), Samsun
- Ukraine (20):
  - COMMUNAL NONPROFIT ENTERPRISE "CLINICAL CENTER OF ONCOLOGY, HEMATOLOGY, TRANSPLANTOLOGY AND PALLIATI ( Site 3671), Cherkasy, Cherkasy Oblast
  - ME І.І. Mechnykov Dnipro Regional Clinical Hospital ( Site 3668), Dnipro, Dnipropetrovsk Oblast
  - Municipal Non-profit Enterprise "City Clinical Hospital #4" of Dnipro City Council ( Site 3650), Dnipro, Dnipropetrovsk Oblast
  - MI Kryvyi Rih Oncology Dispensary of Dnipropetrovsk Regional-Chemotherapy department ( Site 3657), Kryvyi Rih, Dnipropetrovsk Oblast
  - Communal Non-Commercial Enterprise "Prykarpatski Clinical Oncological Center" of Ivano-Frankivsk Reg ( Site 3663), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - MNPE Regional Center of Oncology ( Site 3665), Kharkiv, Kharkivs’ka Oblast’
  - SO"Grigoriev Inst for Med Radiolgy and Oncology of NAMS of Ukraine" ( Site 3666), Kharlkiv, Kharkivs’ka Oblast’
  - Private Enterprise Private Manufacturing Company Acinus-Medical and Diagnostic Centre ( Site 3656), Kropyvnytskyi, Kirovohrad Oblast
  - Asklepion Medical Center ( Site 3667), Khodosovka, Kyivska Oblast
  - National Cancer Institute-Department of Minimally Invasive and Endoscopic Surgery, Interventional R ( Site 3658), Kyiv, Kyivska Oblast
  - LLC Clinic Verum Expert ( Site 3669), Kyiv, Kyivska Oblast
  - Municipal non-profit enterprise "Kyiv City Clinical Oncology Center" of executive body of Kyiv City ( Site 3651), Kyiv, Kyivska Oblast
  - Municipal institution of Lviv regional council Lviv Oncology-Chemotherapy ( Site 3653), Lviv, Lviv Oblast
  - Odessa Regional Oncology Center ( Site 3655), Odesa, Odesa Oblast
  - Sumy regional clinical oncological dispensary-Oncothoracic department ( Site 3661), Sumy, Sumska Oblast
  - Communal Noncommercial Enterprise "Podillia Regional Oncology Center Of Vinnytsia Regional Council" ( Site 3662), Vinnytsia, Vinnytsia Oblast
  - Transcarpathian Regional Clinical Oncology Center-Chemotherapy dept. ( Site 3652), Uzhhorod, Zakarpattia Oblast
  - Uzhhorod City Multidisciplinary Clinical Hospital ( Site 3672), Uzhhorod, Zakarpattia Oblast
  - Municipal non-profit enterprise "Zaporizhzhia regional clinical hospital" of Zaporizhzhia regional c ( Site 3664), Zaporizhzhia, Zaporizhzhia Oblast
  - Zhytomyr Regional Oncology Center ( Site 3670), Zhytomyr, Zhytomyr Oblast
- United Kingdom (19):
  - Aberdeen Royal Infirmary-Department of Oncology ( Site 0521), Aberdeen, Aberdeen City
  - Addenbrookes Hospital ( Site 0522), Cambridge, Cambridgeshire
  - Western General Hospital ( Site 0502), Edinburgh, Edinburgh, City of
  - The Christie ( Site 0516), Manchester, England
  - Weston Park Hospital ( Site 0519), Sheffield, England
  - Mid Essex Hospitals Service Trust. Broomfield Hospital ( Site 0503), Broomfield, Essex
  - The Beatson West of Scotland Cancer Centre ( Site 0506), Glasgow, Glasgow City
  - Royal Preston Hospital ( Site 0518), Preston, Lancashire
  - Barts Health NHS Trust ( Site 0512), London, London, City of
  - University College London Hospital-Cancer Clinical Trials Unit ( Site 0520), London, London, City of
  - Royal Free Hospital ( Site 0507), London, London, City of
  - Royal Marsden Hospital ( Site 0505), London, London, City of
  - Sarah Cannon Research UK ( Site 0504), London, London, City of
  - Belfast City Hospital ( Site 0508), Belfast, Northern Ireland
  - Nottingham University Hospitals NHS Trust ( Site 0510), Nottingham, Nottinghamshire
  - University Hospital Coventry & Warwickshire ( Site 0524), Coventry
  - St James University Hospital ( Site 0509), Leeds
  - The Royal Marsden NHS Foundation Trust. ( Site 0513), Sutton
  - New Cross Hospital-Department of Oncology ( Site 0517), Wolverhampton
- Vietnam (3):
  - Hanoi Oncology Hospital ( Site 3780), Hanoi, Hanoi
  - K Hospital - National Cancer Hospital ( Site 3783), Hanoi, Hanoi
  - National Lung Hospital ( Site 3781), Hanoi, Hanoi

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Robert C, Carlino MS, McNeil C, Ribas A, Grob JJ, Schachter J, Nyakas M, Kee D, Petrella TM, Blaustein A, Lotem M, Arance A, Daud AI, Hamid O, Larkin J, Anderson J, Krepler C, Grebennik D, Long GV. Seven-Year Follow-Up of the Phase III KEYNOTE-006 Study: Pembrolizumab Versus Ipilimumab in Advanced Melanoma. J Clin Oncol. 2023 Aug 20;41(24):3998-4003. doi: 10.1200/JCO.22.01599. Epub 2023 Jun 22. PMID 37348035
- [Result] Long GV, Carlino MS, McNeil C, Ribas A, Gaudy-Marqueste C, Schachter J, Nyakas M, Kee D, Petrella TM, Blaustein A, Lotem M, Arance AM, Daud AI, Hamid O, Larkin J, Yao L, Singh R, Lal R, Robert C. Pembrolizumab versus ipilimumab for advanced melanoma: 10-year follow-up of the phase III KEYNOTE-006 study. Ann Oncol. 2024 Dec;35(12):1191-1199. doi: 10.1016/j.annonc.2024.08.2330. Epub 2024 Sep 15. PMID 39306585
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26277&tenant=MT_MSD_9011